CLINICAL TRIAL: NCT01164462
Title: Feasibility and Limitations of Offering Community Based Rapid HIV Testing to Men Who Have Sex With Men (MSM)
Acronym: DRAG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: French National Agency for Research on AIDS and Viral Hepatitis (Other Government)
Responsible Party: Sponsor
Organization: ANRS, Emerging Infectious Diseases (Other Government)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: AO00439-48
Record Dates: First submitted 2010-07-15; First posted 2010-07-16 (Estimated); Last update posted 2012-12-27 (Estimated); Status verified 2012-12

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- A 2 (Other): During the normal opening hours of five testing centers, clients with a rapid finger-stick blood specimen test
  Interventions: Biological: blood test: rapid finger-stick blood specimen test; Biological: blood test: conventional test
- B group (Other): During evenings and week-ends (i.e. when the centers are closed) only community based with rapid HIV testing
  Interventions: Biological: blood test: rapid finger-stick blood specimen test; Biological: blood test: conventional test
- A1 group (Other): During the normal opening hours of five testing centers, clients with a conventional test.
  Interventions: Biological: blood test: conventional test

INTERVENTIONS:
Biological: blood test: rapid finger-stick blood specimen test
  Arms: A 2; B group
Biological: blood test: conventional test

SUMMARY:
Objective: This research agreement brings together French and Canadian teams of scientists, HIV testing centers and community based partners. The aim is to explore the feasibility and limitations of offering community based rapid HIV testing to men who have sex with men (MSM).

DETAILED DESCRIPTION:
Background: Studies have shown that knowing one's own HIV positive status, may lead to a reduction in sexual risk behaviours. The introduction of new forms of rapid HIV testing in urban areas, may be of benefit to the public health sector, notably in identifying primary HIV infection, preventing secondary HIV transmission and decreasing the spread of HIV infection. Studies have also shown that rapid HIV testing, which yields same-day results, enables a greater number of individuals in populations at risk to become aware of their HIV status.

Issue: The working hypothesis is that the current screening system is not sufficiently suitable for MSM. A community-based rapid HIV testing program could better target the high risk MSM population and shorten the delay between risky behaviour and HIV testing.

Design: This intervention could enable the assessment of the feasibility of community-based rapid HIV testing. Moreover it could compare traditional CDAG (Free Anonymous Screening Consultation or Centre de dépistage anonyme et gratuit in French) center testing with community-based rapid testing. A pre-study phase is first realised to characterize those in the MSM population undergoing HIV testing, before promoting and then beginning the survey. During the normal opening hours of five testing centers, clients will be randomized to have a rapid finger-stick blood specimen test or a conventional test. During evenings and week-ends (i.e. when the centers are closed) only community based rapid HIV testing will be proposed.

Schedule: The pre-study phase is planned for the first quarter of 2009. Promotion of the survey will begin one month before the experimental study which in turn will start in the third quarter of 2009 and will run for 7 months. The end of data analyses is planned for the end of 2010.

Outcome: We will compare HIV population exposure, screening history and the frequency of primary HIV infection diagnosis. We expect to find that those MSM who undergo community based HIV testing during evenings or week-ends, is a population who take repeated sexual risks and who have repeated HIV testing. We also expect to find that this form of testing will be characterized in terms of satisfaction as non-inferior compared to the classic one. In the long term, and if the results are confirmed, rapid HIV testing could be extended to strictly community-based sites.

ELIGIBILITY:
Inclusion Criteria:

* men who have sex with men
* Age ≥ 18 years
* Able to give written consent
* able to give written authorization for lifting anonymity if there is doubt of results
* Covered by French Social Security

Exclusion Criteria:

* who have had a previous diagnosis of seropositivity
* treated by antiretroviral
* woman

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 357 (Actual)
Dates: Start 2010-03; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
the feasibility of community-based rapid HIV testing. testing with community-based rapid testing

SECONDARY OUTCOMES:
Moreover it could compare traditional CDAG (Free Anonymous Screening Consultation) center

CONTACTS AND LOCATIONS:
Overall Officials: Vernay Vaisse Chantal, Principal Investigator — DGAS DPMIS Marseille
Locations (3):
- France (3):
  - CDAG (Free Anonymous Screening Consultation) center, Marseille
  - CDAG (Free Anonymous Screening Consultation) center, Nice
  - CDAG (Free Anonymous Screening Consultation) center, Paris

REFERENCES:
- See also: ((legal sponsor's website)) — http://anrs.fr